CLINICAL TRIAL: NCT02634840
Title: A Modified Technique of Mandibular Ramus Sagittal Split Osteotomy for Prevention of Inferior Alveolar Nerve Injury: A Prospective Cohort Study and Outcome Assessment
Brief Title: Assessment of Nerve Function After Mandible Surgery With a Modified Bilateral Sagittal Split Osteotomy Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG381601-3; CGMH-IRB-101-5264B (Other: CGMH-IRB)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Neurosensory Function of Inferior Alveolar Nerve
Keywords: inferior alveolar nerve; neurosensory disturbance; bilateral sagittal spilt osteotomy; mandibular surgery; neurosensory function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical intervention (Experimental): Patients receiving our modified bilateral sagittal split osteotomy procedure during orthognathic surgery, "intervention arm" in prospective cohort study
  Interventions: Procedure: bilateral sagittal split osteotomy

INTERVENTIONS:
Procedure: bilateral sagittal split osteotomy — surgical technique to split the mandibular ramus through three osteotomy lines on the medial-cranial, buccal-caudal and anterior surface to facilitate a split of the posterior border of the mandible without injury of the inferior alveolar nerve
  Other Names: bilateral ramus sagittal split osteotomy

SUMMARY:
Several technical modifications based on the anatomical position of the neurovascular bundle and its bony mandibular canal have been developed, aiming to prevent injury to the intraalveolar nerve We hypothesized that the incidence of neurosensory disturbance (NSD) should be reduced using our bilateral sagittal split osteotomy (BSSO) technique, because direct intra-alveolar nerve injury can be avoided. The aim of this study was to introduce our modified BSSO technique and evaluate the subsequent incidence of postoperative neurosensory disturbance of the IAN.

DETAILED DESCRIPTION:
The study was designed as a prospective cohort study. Consecutive patients scheduled for orthognathic surgery (OGS) conducted by the senior author at the Craniofacial Center, Department of Plastic and Reconstructive Surgery, Chang Gung Memorial Hospital between January and August 2013 were asked to participate. OGS procedures included mandibular BSSO with or without maxillary LeFort I osteotomy or genioplasty. Fifty-seven patients were enrolled. All patients received cone-beam computed tomography before surgery for intra-alveolar nerve (IAN) assessment and virtual surgery planning.

During surgery, corticotomy and osteotomy lines are modified from the Obwegeser-Dal Pont method. After corticotomy completion, a Dautrey osteotome is driven into the mandible medulla via the anterior corticotomy, keeping constant contact to the inner side of the buccal ramus cortex for the first 10mm. The osteotome, located anterior and lateral to the IAN, is then twisted with moderate force, gradually separating the proximal and distal segment cortices along the anterior opening to facilitate visualization. Possible resistance to open the cortices indicates incomplete corticotomies located in the medial cortex, or the posterior and inferior aspects of both corticotomy lines. Before the complete split, the IAN is evaluated for any exposure through the anterior opening . If the IAN is exposed or attached to the outer cortex, it can gently be replaced into the distal segment. Under visualization through the anterior opening, a straight 4 or 6 mm osteotome is then inserted lateral to and passed beyond the IAN, and then hit to split the posterior ramus cortex along the inner surface of the proximal segment to reach the posterior border.

A standardized record form was provided to all subjects before and after surgery. Gender, preoperative diagnosis and operative details were collected, including surgical plan, mandibular movement extent and concomitant surgical procedures i.e. LeFort I and genioplasty, problematic mandibular splitting and type of fixation. All BSSO procedures were divided into independent left and right sides. After successful splitting of the mandibular ramus, splitting results were categorized.

A 5-point scale self-assessment questionnaire was used during the routine follow up visits to evaluate IAN neurosensory disturbance (NSD) after the BSSO procedure. The subjective neurosensory status evaluation was performed preoperatively, one week, 6 and 12 months postoperatively or until normal sensation returned.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving mandibular bilateral sagittal split osteotomy during orthognathic surgery with normal preoperative intraalveolar nerve function
* patients with cleft lip/palate or hemifacial microsomia were also included

Exclusion Criteria:

* craniofacial syndromic condition, abnormal psychomotor development or previous history of mandibular fracture

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of NSD 12 months postoperatively in relation to IAN exposure during surgery | preoperative to at least 12 months after surgery or return of normal sensation; if no return of normal sensation, reevaluation after another 3 months with computer tomography and clinical exam
  For every patient, the incidence of IAN exposure is recorded. The incidence of NSD is evaluated 12 months after the procedure. The relation and statistical significance is documented with Chi-square-test.

SECONDARY OUTCOMES:
Longitudinal incidence of NSD in relation to gender, age, affected side, preexisting deformity, third molar extraction and genioplasty | preoperative to at least 12 months after surgery or return of normal sensation; if no return of normal sensation, reevaluation after another 3 months with computer tomography and clinical exam
  Subanalysis of the patients in the above mentioned fashion. Clinical evaluation of neurosensory disturbance level of the intraalveolar nerve is carried out with self-assessment questionnaire grading as 1. Affected mandibular side is completely numb, 2. Affected mandibular side is numb with almost no sensation, 3. Affected mandibular side sensation is reduced with some intact sensation, 4. Affected mandibular side has almost normal sensation, 5. Completely normal sensation, no change at all. Subjective neurosensory status evaluation is performed preoperatively, one week, 6 and 12 months postoperatively or until normal sensation return, and absence of neurosensory disturbance was defined with the cutoff at 5 points in the scale. Neurosensory disturbance scores of 1 to 4 are considered abnormal. If the disturbance persists over 12 months, computed tomography and clinical evaluation are performed after additional 3 months.
Longitudinal incidence of NSD in relation to split type during surgery | preoperative to at least 12 months after surgery or return of normal sensation; if no return of normal sensation, reevaluation after another 3 months with computer tomography and clinical exam
  Subanalysis of the patients in the above mentioned fashion. After blinding and light touch on the areas with an 18 gauge needle, participants were asked to choose a score for each one of the tested sites from a scale of 1 to 5. The lowest score was rated as the neurosensory status score at the time of evaluation. Subjective neurosensory status evaluation is performed preoperatively, one week, 6 and 12 months postoperatively or until normal sensation return, and absence of neurosensory disturbance was defined with the cutoff at 5 points in the scale. Neurosensory disturbance scores of 1 to 4 are considered abnormal. If the disturbance persists over 12 months, computed tomography and clinical evaluation are performed after additional 3 months.
Longitudinal incidence of NSD in relation to IAN exposure | preoperative to at least 12 months after surgery or return of normal sensation; if no return of normal sensation, reevaluation after another 3 months with computer tomography and clinical exam
  Subanalysis of the patients in the above mentioned fashion. After blinding and light touch on the areas with an 18 gauge needle, participants were asked to choose a score for each one of the tested sites from a scale of 1 to 5. The lowest score was rated as the neurosensory status score at the time of evaluation. Subjective neurosensory status evaluation is performed preoperatively, one week, 6 and 12 months postoperatively or until normal sensation return, and absence of neurosensory disturbance was defined with the cutoff at 5 points in the scale. Neurosensory disturbance scores of 1 to 4 are considered abnormal. If the disturbance persists over 12 months, computed tomography and clinical evaluation are performed after additional 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lun-Jou Lo, MD, Study Director — Chairman, Department of Surgery, Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obwegeser HL. Orthognathic surgery and a tale of how three procedures came to be: a letter to the next generations of surgeons. Clin Plast Surg. 2007 Jul;34(3):331-55. doi: 10.1016/j.cps.2007.05.014. PMID 17692696
- [Background] Westermark A, Bystedt H, von Konow L. Inferior alveolar nerve function after sagittal split osteotomy of the mandible: correlation with degree of intraoperative nerve encounter and other variables in 496 operations. Br J Oral Maxillofac Surg. 1998 Dec;36(6):429-33. doi: 10.1016/s0266-4356(98)90458-2. PMID 9881784
- [Background] Ylikontiola L, Kinnunen J, Oikarinen K. Factors affecting neurosensory disturbance after mandibular bilateral sagittal split osteotomy. J Oral Maxillofac Surg. 2000 Nov;58(11):1234-9; discussion 1239-40. doi: 10.1053/joms.2000.16621. PMID 11078134
- [Background] Kane AA, Lo LJ, Chen YR, Hsu KH, Noordhoff MS. The course of the inferior alveolar nerve in the normal human mandibular ramus and in patients presenting for cosmetic reduction of the mandibular angles. Plast Reconstr Surg. 2000 Oct;106(5):1162-74; discussion 1175-6. doi: 10.1097/00006534-200010000-00029. PMID 11039388
- [Background] Hanzelka T, Foltan R, Pavlikova G, Horka E, Sedy J. The role of intraoperative positioning of the inferior alveolar nerve on postoperative paresthesia after bilateral sagittal split osteotomy of the mandible: prospective clinical study. Int J Oral Maxillofac Surg. 2011 Sep;40(9):901-6. doi: 10.1016/j.ijom.2011.04.002. Epub 2011 May 13. PMID 21570811
- [Background] Colella G, Cannavale R, Vicidomini A, Lanza A. Neurosensory disturbance of the inferior alveolar nerve after bilateral sagittal split osteotomy: a systematic review. J Oral Maxillofac Surg. 2007 Sep;65(9):1707-15. doi: 10.1016/j.joms.2007.05.009. PMID 17719387
- [Background] Agbaje JO, Salem AS, Lambrichts I, Jacobs R, Politis C. Systematic review of the incidence of inferior alveolar nerve injury in bilateral sagittal split osteotomy and the assessment of neurosensory disturbances. Int J Oral Maxillofac Surg. 2015 Apr;44(4):447-51. doi: 10.1016/j.ijom.2014.11.010. Epub 2014 Dec 9. PMID 25496848